CLINICAL TRIAL: NCT00056368
Title: A Phase III, Double-Blind, Randomized, Multi-Center, Study of the Safety and Efficacy of Anidulafungin vs. Fluconazole in the Treatment of Patients With Candidemia and Other Forms of Invasive Candidiasis and Prevention of Complications.
Brief Title: The Safety and Efficacy of Anidulafungin Versus Comparator in Patients With Candidemia and Invasive Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Vicuron Pharmaceuticals (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VER002-9; A8851002
Record Dates: First submitted 2003-03-11; First posted 2003-03-12 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Candidiasis
Keywords: Candida blood stream infections; Candida infections; Candidemia; Invasive Candidiasis
MeSH Terms: conditions — Candidiasis; Candidemia; Candidiasis, Invasive | interventions — Anidulafungin; Fluconazole

INTERVENTIONS:
Drug: Anidulafungin
Drug: Fluconazole

SUMMARY:
Anidulafungin is a medicine being developed for treatment of patients with certain kinds of fungal infections. These infections due to yeast (a type of fungus) in the mouth/esophagus, in the blood or in other areas within the body.

DETAILED DESCRIPTION:
Anidulafungin is an investigational drug being developed as an intravenous treatment for esophageal candidiasis, candidemia and other invasive fungal infections. Anidulafungin is an antifungal agent of the echinocandin class, which targets the fungal cell wall of yeast and other filamentous fungi.

ELIGIBILITY:
* Diagnosis of candidemia and/or other forms of invasive candidiasis.
* Should not have received greater than 48 hours of systemic antifungal therapy.
* Life expectancy should be greater than 72 hours.
* Should not have received greater than one week of prophylactic azole therapy 30 days prior to enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2003-03; Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Versicor, Inc., King of Prussia, Pennsylvania, United States

REFERENCES:
- [Derived] Reboli AC, Rotstein C, Pappas PG, Chapman SW, Kett DH, Kumar D, Betts R, Wible M, Goldstein BP, Schranz J, Krause DS, Walsh TJ; Anidulafungin Study Group. Anidulafungin versus fluconazole for invasive candidiasis. N Engl J Med. 2007 Jun 14;356(24):2472-82. doi: 10.1056/NEJMoa066906. PMID 17568028